CLINICAL TRIAL: NCT04496687
Title: The International Spontaneous Coronary Artery Dissection "iSCAD" Registry (SCAD)
Brief Title: International Spontaneous Coronary Artery Dissection (SCAD) "iSCAD" Registry
Status: Recruiting | Type: Observational
Sponsor: SCAD Alliance (Other)
Collaborators: PERFUSE Study Group (Unknown)
Responsible Party: Sponsor
Other Study IDs: 20190308
Record Dates: First submitted 2020-07-29; First posted 2020-08-03 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Spontaneous Coronary Artery Dissection
Keywords: spontaneous coronary artery dissection (SCAD); myocardial infarction; sudden cardiac arrest; acute coronary syndrome
MeSH Terms: conditions — Coronary Artery Dissection, Spontaneous; Myocardial Infarction; Death, Sudden, Cardiac; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of "iSCAD," the International Spontaneous Coronary Artery Dissection (SCAD) Registry, is to serve as an internationally collaborative, multicenter registry coordinated by an experienced and centralized coordinating center in an effort to increase the pace of participant recruitment, and thereby increase statistical power of studies related to SCAD.

The ultimate goal of iSCAD Registry is to facilitate the development of best practices and clinical guidelines for preventing SCAD or its recurrence. This observational study will be prospective and retrospective in its recruitment and will collect clinical information to better understand the natural history and prognosis for SCAD.

DETAILED DESCRIPTION:
Spontaneous Coronary Artery Dissection (SCAD) is an under-diagnosed cause of acute coronary syndrome (ACS), myocardial infarction (MI) and sudden cardiac arrest. The inner lining of the coronary artery splits and allows blood to seep into the adjacent layer, forming a blockage (hematoma), or the artery continues to tear, creating a flap of tissue that blocks blood flow in the artery.

SCAD strikes generally healthy, younger individuals (average age 42) who do not have traditional cardiac risk factors. Warning signs of SCAD encompass the full range of ACS and MI symptoms, from vague to classic. The cause of SCAD is currently unknown and the psychosocial impact of SCAD is traumatizing. The work of the iSCAD Registry will encompass the physical and psychosocial study of SCAD.

ELIGIBILITY:
Inclusion Criteria:

Participants with a new diagnosis of SCAD or a history of confirmed or suspected SCAD will be prospectively recruited from either:

1. Inpatient wards of the enrolling medical centers during the acute presentation of SCAD, or
2. Outpatient cardiovascular clinics of enrolling medical centers.

Participants must be:

* 18 years of age or older
* Diagnosis of SCAD or history of SCAD based on coronary angiography, either catheter-based or coronary CTA
* Suspected SCAD by coronary angiography

Exclusion Criteria:

1. Coronary dissection in association with atherosclerosis or as a result of iatrogenic injury
2. Inability to provide informed consent
3. Inability to complete study-related patient questionnaires
4. Inability to understand and complete patient questionnaires independently

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Spontaneous coronary artery dissection (SCAD) is defined as the non-traumatic, non-iatrogenic separation of the coronary arterial wall by intramural hemorrhage creating a false lumen, with or without an intimal tear. SCAD nearly always presents as an acute myocardial infarction. The prevalence of SCAD varies depending on the population studied. A goal of iSCAD Registry is to expand diversity of race, ethnicity, and sex of study participants. The mean age of SCAD presentation is 45-53 years of age, and appears to primarily affect women.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-03-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Descriptive Data | Continuous time frame following index event for an average of 3 years from study contact date
  Participant demographic, historical, clinical characteristics, and treatment data
Clinical Outcomes | Continuous time frame following index event for an average of 3 years from study contact date
  Prospectively collected long-term outcomes including recurrent myocardial infarction, hospitalization, heart failure, stroke or transient ischemic attack, arrhythmia, and all cause mortality
Psychosocial Outcomes | Continuous time frame following index event for an average of 3 years from study contact date
  Prospectively collected data on participant's mental health using validated questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Esther Kim, MD, Study Chair — Chair, Steering Committee; Malissa Wood, MD, Principal Investigator — Member, Steering Committee; Sahar Naderi, MD, Principal Investigator — Member, Steering Committee
Locations (31):
- United States (30):
  - Cedars Sinai, Los Angeles, California
  - UCLA (University of California, Los Angeles), Los Angeles, California
  - Kaiser Permanente Northern California, San Francisco, California
  - University of Colorado, Aurora, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - University of South Florida, Tampa, Florida
  - Emory Healthcare System, Atlanta, Georgia
  - Northwestern Medicine, Chicago, Illinois
  - University of Kentucky, Lexington, Kentucky
  - Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - St. Luke's Mid America, Kansas City, Missouri
  - Washington University, St Louis, Missouri
  - Dartmouth-Hitchcock, Lebanon, New Hampshire
  - Catholic Medical Center, Manchester, New Hampshire
  - Mount Sinai, New York, New York
  - Columbia University Medical Center, New York, New York
  - Atrium Health Sanger Heart and Vascular Institute, Charlotte, North Carolina
  - University Hospitals--Case Western, Cleveland, Ohio
  - Oklahoma Heart, Oklahoma City, Oklahoma
  - Providence, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Allegheny Health Network, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UT Southwestern, Dallas, Texas
  - Intermountain, Murray, Utah
  - University of Virginia, Charlottesville, Virginia
  - Inova Heart & Vascular Institute, Fairfax, Virginia
  - University of Washington Medicine, Seattle, Washington
- Victor Chang Cardiac Research Institute, Darlinghurst, New South Wales, Australia

REFERENCES:
- [Derived] Sumner JA, Kim ESH, Wood MJ, Chi G, Nolen J, Grodzinsky A, Gornik HL, Kadian-Dodov D, Wells BJ, Hess CN, Lewey J, Tam L, Henkin S, Orford J, Wells G, Kumbhani DJ, Lindley KJ, Gibson CM, Leon KK, Naderi S. Posttraumatic Stress Disorder After Spontaneous Coronary Artery Dissection: A Report of the International Spontaneous Coronary Artery Dissection Registry. J Am Heart Assoc. 2024 Apr 2;13(7):e032819. doi: 10.1161/JAHA.123.032819. Epub 2024 Mar 27. PMID 38533943
- See also: iSCAD Registry Home Page — https://iscadregistry.bidmc.org/index.php/Main_Page
- See also: iSCAD Registry FAQs and sponsor page — https://www.scadalliance.org/iscad-registry/